CLINICAL TRIAL: NCT00881816
Title: Phase I Clinical Study of Liposomal Paclitaxel Plus Capecitabine in Chinese Patients With Advanced Gastric Carcinoma
Brief Title: Dose Escalation Study of Liposomal Paclitaxel Plus Capecitabine in Chinese Patients With Advanced Gastric Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Dr. Li Jin, Cancer Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS-GC-02-2008; NJSK-LPS-PH I-02
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Advanced Gastric Carcinoma
Keywords: Liposomal Paclitaxel; Capecitabine; Maximum tolerated dose; Dose limiting toxicity
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposomal paclitaxel plus capecitabine (Experimental)
  Interventions: Drug: Liposomal paclitaxel plus capecitabine

INTERVENTIONS:
Drug: Liposomal paclitaxel plus capecitabine — All Patients will receive liposomal paclitaxel (with a dose of 60mg/m2,3h,ivgtt,at d1,8,15) and capecitabine (with a dose of 1600mg/m2,bid,po.,at d1-14),each cycle for 4 cycles.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and dose limiting toxicity of liposomal paclitaxel plus capecitabine in Chinese patients with advanced gastric carcinoma.

DETAILED DESCRIPTION:
There are clinical trials showed that taxane is optional for the treatment of gastric cancer. Liposomal paclitaxel has different pharmacokinetic features comparing with conventional taxane. This study is designed to find the maximum tolerated dose and dose limiting toxicity of liposomal paclitaxel combined with capecitabine in Chinese patients with advanced gastric carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75
* Histologically or cytologically documented gastric adenocarcinoma and esophagus-gastro adenocarcinoma of metastatic or advanced stages with/without measurable tumor according to RECIST standard
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Patients who are expected to live at least 3 months
* No prior systemic chemotherapy with advanced stereo- tumor before the recruitment(recidivist/ metastatic without perioperative chemotherapy at least 6m)
* No Previous anaphylactic reaction to hormone
* Obtaining informed consent
* Patients may comply with the study protocol
* Laboratory tests: Absolute neutrophil count (ANC) ≥2,000/mm³, Platelet count ≥100,000/mm³, Hemoglobin ≥9.0 g/dL, Serum creatinine≤1.5 x the institutional upper limit of normal (ULN), Creatinine clearance≥50ml/min，Total bilirubin≤1.5 x the institutional upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 x ULN. In the case of known liver metastasis, ALT and AST（SGOT） ≤1.5 x ULN.

Exclusion Criteria:

* Active uncontrolled central nervous system metastasis
* No adequate organ function or known disease :

  * myocardial infarction
  * active heart disease
  * neuropathy or mental diseases including dementia or epilepsy
  * blind、deaf、dumb or extremity disability
  * known infection
  * active diffuse intravascular coagulation
  * known infection with hepatitis virus
* Pregnant or nursing,fertile patients would not use effective contraception during study treatment
* Prior clinically significant gastrointestinal tract disease , that would influence obviously capecitabine to absorb,including the ability to swallow by the attending physician
* No other active malignancies except that in complete remission with squamous cell carcinoma in situ of the cervix or anus, completely resected basal cell carcinoma, or no recrudescence for at least 2 year from the time a response was first documented
* Having other study medication within 4w
* Having radiation therapy or operation within 4w
* Any non-remission toxicity ≥ CTC 1 in prior anticancer therapy(including radiation therapy) (except alopecie and hemoglobin)
* Peripheral nerve disease ≥ 2
* Previous anaphylactic reaction to Capecitabine and Paclitaxel or diluents bases
* Absence of dihydropyrimidine dehydrogenase
* Patients not suitable determined by the attending physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | 6 months

SECONDARY OUTCOMES:
dose limiting toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Dr., Principal Investigator — Cancer Hospital of Fudan University